CLINICAL TRIAL: NCT03104374
Title: A Phase 3, Randomized, Double-Blind, Study Comparing Upadacitinib (ABT-494) to Placebo in Subjects With Active Psoriatic Arthritis Who Have a History of Inadequate Response to at Least One Biologic Disease Modifying Anti-Rheumatic Drug (bDMARD)
Brief Title: A Study Comparing Upadacitinib (ABT-494) to Placebo in Participants With Active Psoriatic Arthritis Who Have a History of Inadequate Response to at Least One Biologic Disease Modifying Anti-Rheumatic Drug
Acronym: SELECT - PsA 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-554; 2016-004152-30 (EudraCT Number)
Record Dates: First submitted 2017-04-04; First posted 2017-04-07 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Psoriatic Arthritis
Keywords: Arthritis; Psoriasis; Anti-Rheumatic; Anti-inflammatory; Joint disease; Musculoskeletal disease
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Psoriasis; Joint Diseases; Musculoskeletal Diseases | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Upadacitinib 15 mg (Experimental): Administered once daily.
  Interventions: Drug: Upadacitinib
- Placebo / Upadacitinib 30 mg (Placebo Comparator): Administered once daily.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- Upadacitinib 30 mg (Experimental): Administered once daily.
  Interventions: Drug: Upadacitinib
- Placebo / Upadacitinib 15 mg (Placebo Comparator): Administered once daily.
  Interventions: Drug: Placebo; Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Oral tablet
  Arms: Placebo / Upadacitinib 15 mg; Placebo / Upadacitinib 30 mg
Drug: Upadacitinib — Oral tablet
  Other Names: ABT-494

SUMMARY:
This is a Phase 3 multicenter study that included two periods. Period 1 was designed to compare the safety, tolerability, and efficacy of upadacitinib 15 mg once daily (QD) and 30 mg QD versus placebo in participants with moderately to severely active Psoriatic Arthritis (PsA) who had an inadequate response to Biological Disease Modifying Anti-Rheumatic Drug (bDMARDs). Period 2 evaluated the safety, tolerability and efficacy of upadacitinib 15 mg QD and 30 mg QD in subjects with PsA who completed Period 1.

DETAILED DESCRIPTION:
The study included a 35-day screening period; a 56-week blinded period which included 24 weeks of randomized, double-blind, parallel-group, placebo-controlled treatment followed by an additional 32 weeks of treatment blinded to the dose of upadacitinib (Period 1); a long-term extension period of up to a total treatment duration of up to approximately 3 years (Period 2); and a 30-day follow-up call or visit.

All participants in Period 1 who were randomized to receive Placebo up to 24 weeks were pooled for the assessment of all outcome measures. All participants receiving upadacitinib 30 mg QD during Period 2 were switched to upadacitinib 15 mg QD following a protocol amendment and were pooled for AE reporting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PsA with symptom onset at least 6 months prior to the Screening Visit and fulfillment of the Classification Criteria for PsA (CASPAR) criteria
* Participant has active disease at Baseline defined as >= 3 tender joints (based on 68 joint counts) and >= 3 swollen joints (based on 66 joint counts) at Screening and Baseline Visits
* Diagnosis of active plaque psoriasis or documented history of plaque psoriasis
* Participant has had an inadequate response (lack of efficacy after a minimum 12 week duration of therapy) or intolerance to treatment with at least 1 bDMARD.

Exclusion Criteria:

* Prior exposure to any Janus Kinase (JAK) inhibitor (including but not limited to ruxolitinib, tofacitinib, baricitinib, and filgotinib)
* Current treatment with > 2 non-biologic DMARDs or use of DMARDs other than Methotrexate (MTX), Sulfasalazine (SSZ), Leflunomide (LEF), apremilast, Hydroxychloroquine (HCQ), bucillamine or iguratimod or use of MTX in combination with LEF at Baseline.
* History of fibromyalgia, any arthritis with onset prior to age 17 years, or current diagnosis of inflammatory joint disease other than PsA (including, but not limited to rheumatoid arthritis, gout, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, systemic lupus erythematosus). Prior history of reactive arthritis or axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial spondyloarthritis is permitted if documentation of change in diagnosis to PsA or additional diagnosis of PsA is made. Prior history of fibromyalgia is permitted if documentation of change in diagnosis to PsA or documentation that the diagnosis of fibromyalgia was made incorrectly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (165):
- United States (72):
  - Alabama Medical Group, PC /ID# 159836, Mobile, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 160047, Mesa, Arizona
  - Sun Valley Arthritis Center Ltd. /ID# 161203, Peoria, Arizona
  - Duplicate_AZ Arthritis and Rheumotology Research, PLLC /ID# 160006, Phoenix, Arizona
  - Osteoporosis Medical Center /ID# 161411, Beverly Hills, California
  - Covina Arthritis Clinic /ID# 159919, Covina, California
  - Triwest Research Associates /ID# 159915, El Cajon, California
  - Duplicate_Providence Medical Foundation /ID# 160005, Fullerton, California
  - C.V. Mehta MD, Med Corporation /ID# 161192, Hemet, California
  - Care Access Research, Huntington Beach /ID# 160049, Huntington Beach, California
  - Purushotham & Akther Kotha MD, Inc /ID# 159834, La Mesa, California
  - Stanford University School of Med /ID# 161402, Stanford, California
  - Inland Rheum Clin Trials Inc. /ID# 159839, Upland, California
  - Medvin Clinical Research /ID# 160045, Whittier, California
  - Denver Arthritis Clinic /ID# 159899, Denver, Colorado
  - Colorado Arthritis Associates /ID# 159856, Lakewood, Colorado
  - Duplicate_Arthritis & Rheumatic Disease Specialties /ID# 161409, Aventura, Florida
  - International Medical Research /ID# 160051, Daytona Beach, Florida
  - Precision Research Organization /ID# 161293, Miami Lakes, Florida
  - Duplicate_Suncoast Clinical Research /ID# 161417, New Port Richey, Florida
  - Millennium Research /ID# 159833, Ormond Beach, Florida
  - Arthritis Center, Inc. /ID# 163463, Palm Harbor, Florida
  - Gulf Region Clinical Res Inst /ID# 159860, Pensacola, Florida
  - Sarasota Arthritis Center /ID# 159854, Sarasota, Florida
  - BayCare Medical Group /ID# 161405, St. Petersburg, Florida
  - West Broward Rheumatology Associates /ID# 161412, Tamarac, Florida
  - Clinical Research of West Florida - Tampa /ID# 160069, Tampa, Florida
  - Clinical Research of West Florida, Inc /ID# 159840, Tampa, Florida
  - USF Health Morsani Center for /ID# 161291, Tampa, Florida
  - BayCare Medical Group, Inc. /ID# 159912, Tampa, Florida
  - Florida Medical Clinic /ID# 160013, Zephyrhills, Florida
  - Jefrey D. Lieberman, MD, P.C. /ID# 159842, Decatur, Georgia
  - Atlanta Research Center for Rheumatology /ID# 161201, Marietta, Georgia
  - Velocity Clinical Research - Boise /ID# 159922, Meridian, Idaho
  - Great Lakes Clinical Trials /ID# 163438, Chicago, Illinois
  - Deerbrook Medical Associates /ID# 159815, Libertyville, Illinois
  - Duplicate_Clinic of Robert Hozman/Clinical Investigation Specialists /ID# 160068, Skokie, Illinois
  - The Arthritis & Diabetes Clinic, Inc. /ID# 161294, Monroe, Louisiana
  - Arthritis Treatment Center /ID# 160053, Frederick, Maryland
  - The Center for Rheumatology and Bone Research /ID# 159900, Wheaton, Maryland
  - Clinical Pharmacology Study Group /ID# 158712, Worcester, Massachusetts
  - Clinvest Research LLC /ID# 161208, Springfield, Missouri
  - Westroads Clinical Research /ID# 160004, Omaha, Nebraska
  - Atlantic Coast Research /ID# 159810, Toms River, New Jersey
  - Duplicate_Arthritis and Osteo Assoc /ID# 160015, Las Cruces, New Mexico
  - Center for Rheumatology LLP /ID# 167046, Albany, New York
  - St. Lawrence Health System /ID# 159857, Potsdam, New York
  - DJL Clinical Research, PLLC /ID# 161414, Charlotte, North Carolina
  - Physicians East, PA /ID# 159898, Greenville, North Carolina
  - Shanahan Rheuma & Immuno /ID# 160012, Raleigh, North Carolina
  - PMG Research of Wilmington LLC /ID# 161403, Wilmington, North Carolina
  - Trinity Health Med Arts Clinic /ID# 159811, Minot, North Dakota
  - STAT Research, Inc. /ID# 161416, Vandalia, Ohio
  - Health Research of Oklahoma /ID# 159913, Oklahoma City, Oklahoma
  - Altoona Ctr Clinical Res /ID# 159861, Duncansville, Pennsylvania
  - University of Pittsburgh MC /ID# 161193, Pittsburgh, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 163462, Summerville, South Carolina
  - Rheumatology Consultants, PLLC /ID# 161408, Knoxville, Tennessee
  - Dr. Ramesh Gupta /ID# 160067, Memphis, Tennessee
  - Tekton Research, Inc. /ID# 160008, Austin, Texas
  - Diagnostic Group /ID# 161406, Beaumont, Texas
  - Arthritis and Osteoporosis Clinic Of Brazos Valley /ID# 163439, College Station, Texas
  - Adriana Pop-Moody MD Clinic PA /ID# 160009, Corpus Christi, Texas
  - Metroplex Clinical Research /ID# 159818, Dallas, Texas
  - Rheumatic Disease Clin Res Ctr /ID# 161252, Houston, Texas
  - Accurate Clinical Research /ID# 160052, Houston, Texas
  - P&I Clinical Research /ID# 159837, Lufkin, Texas
  - SW Rheumatology Res. LLC /ID# 160014, Mesquite, Texas
  - DM Clinical Research - Tomball /ID# 161753, Tomball, Texas
  - Arthritis & Osteoporosis Clinic /ID# 161400, Waco, Texas
  - Arthritis Clinic of N. VA, P.C /ID# 159858, Arlington, Virginia
  - Duplicate_Swedish Medical Center /ID# 159918, Seattle, Washington
- Australia (4):
  - Emeritus Research Sydney /ID# 166751, Botany, New South Wales
  - The Queen Elizabeth Hospital /ID# 200840, Woodville South, South Australia
  - Box Hill Hospital /ID# 166752, Box Hill, Victoria
  - Heidelberg Repatriation Hospital /ID# 167441, Heidelberg West, Victoria
- Belgium (2):
  - ReumaClinic /ID# 164214, Genk, Limburg
  - UZ Gent /ID# 164210, Ghent, Oost-Vlaanderen
- Brazil (7):
  - CIP - Centro Internacional de Pesquisa /ID# 161808, Goiânia, Goiás
  - Faculdade de Medicina do ABC /ID# 163489, Santo André, La Spezia
  - Hospital de Clínicas da Universidade Federal de Uberlândia /ID# 161794, Uberlândia, Minas Gerais
  - Hospital de Clinicas de Porto Alegre /ID# 161795, Porto Alegre, Rio Grande do Sul
  - LMK Sevicos Medicos S/S /ID# 161806, Porto Alegre, Rio Grande do Sul
  - Duplicate_Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 163317, Ribeirão Preto, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 161793, São Paulo
- Canada (5):
  - Percuro Clinical Research, Ltd /ID# 157835, Victoria, British Columbia
  - CIADS Research Co Ltd /ID# 157843, Winnipeg, Manitoba
  - The Waterside Clinic /ID# 157838, Orillia, Ontario
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 157836, Sainte-Foy, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 163557, Trois-Rivières, Quebec
- Chile (4):
  - CTR Estudios Clinicos /ID# 206038, Providencia, Aysén
  - Duplicate_Clinica Dermacross /ID# 169537, Santiago
  - Duplicate_Centro Internacional de Estudios Clinicos /ID# 169543, Santiago
  - Prosalud Ltda. /ID# 169542, Santiago
- Czechia (2):
  - Revmatologie Bruntal, s.r.o /ID# 159632, Prostějov
  - Medical Plus, s.r.o. /ID# 159631, Uherské Hradiště
- France (6):
  - Hopital Saint Joseph /ID# 163755, Marseille, Bouches-du-Rhone
  - CHU Toulouse /ID# 163743, Toulouse, Occitanie
  - Centre Hospitalier du Mans /ID# 163746, Le Mans, Sarthe
  - CHRU Tours - Hopital Trousseau /ID# 163772, Chambray-lès-Tours
  - Duplicate_CHU-Hospital Henri Mondor /ID# 163895, Créteil
  - Duplicate_AP-HP - Hopital Lariboisiere /ID# 163773, Paris
- Greece (3):
  - General Hospital of Athens Laiko /ID# 163474, Athens, Attica
  - Naval Hospital of Athens /ID# 163495, Athens
  - Reg Gen Univ Hosp Larissa /ID# 163493, Larissa
- Hungary (7):
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz /ID# 162573, Győr, Győr-Moson-Sopron
  - Vital Medicina Kft /ID# 162571, Veszprém, Veszprém megye
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 170911, Budapest
  - Revita Reumatologiai Rendelo /ID# 162575, Budapest
  - Obudai Egeszsegugyi Centrum Kft. /ID# 162576, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 162572, Debrecen
  - MÁV Kórház /ID# 162574, Szolnok
- Italy (8):
  - Azienda Ospedaliera Universitaria Federico II /ID# 202410, Napoli, L Aquila
  - Duplicate_Fondazione Policlinico Universitario Campus Bio-Medico di Roma /ID# 164123, Rome, Roma
  - Duplicate_Fondazione PTV Policlinico Tor Vergata /ID# 162749, Rome, Roma
  - Duplicate_Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 162748, Ancona
  - Duplicate_A.O.U. Policlinico G. Rodolico S.Marco- Presidio G.Rodolico /ID# 164126, Catania
  - Duplicate_AOU Arcispedale Sant Anna di /ID# 164127, Cona
  - ASST Gaetano Pini/Presidio Ospedaliero Pini /ID# 164125, Milan
  - Duplicate_Azienda Unita Sanitaria Locale/IRCCS /ID# 162751, Reggio Emilia
- Japan (16):
  - Daido Hospital /ID# 163639, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 162563, Nagoya, Aichi-ken
  - Fukuoka University Hospital /ID# 161774, Fukuoka, Fukuoka
  - Duplicate_Kitakyushu Municipal Medical Center /ID# 163516, Kitakyushu-shi, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan /ID# 161472, Kitakyushu-shi, Fukuoka
  - Asahikawa Medical University Hospital /ID# 200684, Asahikawa-shi, Hokkaido
  - Mie University Hospital /ID# 162085, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 164035, Sendai, Miyagi
  - Oribe Clinic of Rheumatism and Medicine /ID# 163704, Ōita, Oita Prefecture
  - Kansai Medical University Hospital /ID# 162081, Hirakata-shi, Osaka
  - National Hospital Organization Osaka Minami Medical Center /ID# 162589, Kawachinagano Shi, Osaka
  - Osaka Metropolitan University Hospital /ID# 162082, Osaka, Osaka
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 161773, Osaka, Osaka
  - Juntendo University Hospital /ID# 162089, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 162013, Chuo-ku, Tokyo
  - Keio University Hospital /ID# 162130, Shinjuku-ku, Tokyo
- Netherlands (4):
  - Medisch Centrum Leeuwarden /ID# 163049, Leeuwarden, South Holland
  - Duplicate_Erasmus Medisch Centrum /ID# 163052, Rotterdam, South Holland
  - Maasstad Ziekenhuis /ID# 163050, Rotterdam, South Holland
  - Sint Maartenskliniek /ID# 163703, Ubbergen
- New Zealand (4):
  - Duplicate_Middlemore Hospital /ID# 166411, Otahuhu, Auckland
  - Timaru Medical Specialists Ltd /ID# 166410, Timaru, Canterbury
  - Waikato Hospital /ID# 166412, Hamilton, Waikato Region
  - Porter Rheumatology Ltd /ID# 200422, Nelson
- Portugal (5):
  - Duplicate_Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE /ID# 165897, Vila Nova de Gaia, Porto District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 165898, Ponte de Lima, Viana do Castelo District
  - Instituto Portugues De Reumatologia /ID# 165894, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz /ID# 165896, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 165895, Lisbon
- Puerto Rico (3):
  - Alma M. Cruz Santana, MD-Private practice /ID# 163308, Carolina
  - Ponce Medical School Foundation /ID# 163918, Ponce
  - GCM Medical Group PSC /ID# 163716, San Juan
- South Korea (2):
  - Duplicate_Ajou University Hospital /ID# 163893, Suwon, Gyeonggido
  - Duplicate_Inha University Hospital /ID# 163892, Junggu, Incheon Gwang Yeogsi
- Spain (5):
  - Hospital Clinico Universitario Virgen de la Arrixaca /ID# 163138, El Palmar, Murcia
  - Duplicate_Hospital Universitario A Coruna - CHUAC /ID# 161019, A Coruña
  - Duplicate_Hospital Universitario Reina Sofia /ID# 170764, Córdoba
  - Hospital Campus de la Salud /ID# 170768, Granada
  - Hospital Universitario Ramon y Cajal /ID# 161020, Madrid
- United Kingdom (6):
  - Royal United Hospitals Bath /ID# 161054, Bath, Bath And North East Somerset
  - Barts Health NHS Trust /ID# 161053, London, London, City of
  - Guys and St Thomas NHS Foundation Trust /ID# 161063, London, London, City of
  - Duplicate_NHS Greater Glasgow and Clyde /ID# 162712, Glasgow
  - Duplicate_Bedfordshire Hospitals NHS Foundation Trust /ID# 162713, Luton
  - Duplicate_Christchurch University Hospitals Dorset NHS University Hospitals Dors /ID# 162711, Poole

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Burmester GR, Stigler J, Rubbert-Roth A, Tanaka Y, Azevedo VF, Coombs D, Lagunes I, Lippe R, Wung P, Gensler LS. Safety Profile of Upadacitinib up to 5 Years in Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis: An Integrated Analysis of Clinical Trials. Rheumatol Ther. 2024 Jun;11(3):737-753. doi: 10.1007/s40744-024-00671-4. Epub 2024 Apr 29. PMID 38683479
- [Derived] Cantini F, Marchesoni A, Novelli L, Gualberti G, Marando F, McDearmon-Blondell EL, Gao T, McGonagle D, Salvarani C. Effects of upadacitinib on enthesitis in patients with psoriatic arthritis: a post hoc analysis of SELECT-PsA 1 and 2 trials. Rheumatology (Oxford). 2024 Nov 1;63(11):3146-3154. doi: 10.1093/rheumatology/keae057. PMID 38331400
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Mease P, Setty A, Papp K, Van den Bosch F, Tsuji S, Keiserman M, Carter K, Li Y, McCaskill R, McDearmon-Blondell E, Wung P, Tillett W. Upadacitinib in patients with psoriatic arthritis and inadequate response to biologics: 3-year results from the open-label extension of the randomised controlled phase 3 SELECT-PsA 2 study. Clin Exp Rheumatol. 2023 Nov;41(11):2286-2297. doi: 10.55563/clinexprheumatol/8l7bbk. Epub 2023 Jul 5. PMID 37404160
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Mease P, Kavanaugh A, Gladman D, FitzGerald O, Soriano ER, Nash P, Feng D, Lertratanakul A, Douglas K, Lippe R, Gossec L. Disease Control with Upadacitinib in Patients with Psoriatic Arthritis: A Post Hoc Analysis of the Randomized, Placebo-Controlled SELECT-PsA 1 and 2 Phase 3 Trials. Rheumatol Ther. 2022 Aug;9(4):1181-1191. doi: 10.1007/s40744-022-00449-6. Epub 2022 May 23. PMID 35606663
- [Derived] Burmester GR, Winthrop K, Blanco R, Nash P, Goupille P, Azevedo VF, Salvarani C, Rubbert-Roth A, Lesser E, Lippe R, Lertratanakul A, Mccaskill RM, Liu J, Ruderman EM. Safety Profile of Upadacitinib up to 3 Years in Psoriatic Arthritis: An Integrated Analysis of Two Pivotal Phase 3 Trials. Rheumatol Ther. 2022 Apr;9(2):521-539. doi: 10.1007/s40744-021-00410-z. Epub 2021 Dec 30. PMID 34970731
- [Derived] Nash P, Richette P, Gossec L, Marchesoni A, Ritchlin C, Kato K, McDearmon-Blondell EL, Lesser E, McCaskill R, Feng D, Anderson JK, Ruderman EM. Upadacitinib as monotherapy and in combination with non-biologic disease-modifying antirheumatic drugs for psoriatic arthritis. Rheumatology (Oxford). 2022 Aug 3;61(8):3257-3268. doi: 10.1093/rheumatology/keab905. PMID 34864911
- [Derived] Strand V, Van den Bosch F, Ranza R, Leung YY, Drescher E, Zueger P, Saffore CD, Lertratanakul A, Lippe R, Nash P. Patient-Reported Outcomes in Psoriatic Arthritis Patients with an Inadequate Response to Biologic Disease-Modifying Antirheumatic Drugs: SELECT-PsA 2. Rheumatol Ther. 2021 Dec;8(4):1827-1844. doi: 10.1007/s40744-021-00377-x. Epub 2021 Oct 18. PMID 34661885
- [Derived] Muensterman E, Engelhardt B, Gopalakrishnan S, Anderson JK, Mohamed MF. Upadacitinib pharmacokinetics and exposure-response analyses of efficacy and safety in psoriatic arthritis patients - Analyses of phase III clinical trials. Clin Transl Sci. 2022 Jan;15(1):267-278. doi: 10.1111/cts.13146. Epub 2021 Oct 27. PMID 34464029
- [Derived] Mease PJ, Lertratanakul A, Papp KA, van den Bosch FE, Tsuji S, Dokoupilova E, Keiserman MW, Bu X, Chen L, McCaskill RM, Zueger P, McDearmon-Blondell EL, Pangan AL, Tillett W. Upadacitinib in Patients with Psoriatic Arthritis and Inadequate Response to Biologics: 56-Week Data from the Randomized Controlled Phase 3 SELECT-PsA 2 Study. Rheumatol Ther. 2021 Jun;8(2):903-919. doi: 10.1007/s40744-021-00305-z. Epub 2021 Apr 28. PMID 33913086
- [Derived] Mease PJ, Lertratanakul A, Anderson JK, Papp K, Van den Bosch F, Tsuji S, Dokoupilova E, Keiserman M, Wang X, Zhong S, McCaskill RM, Zueger P, Pangan AL, Tillett W. Upadacitinib for psoriatic arthritis refractory to biologics: SELECT-PsA 2. Ann Rheum Dis. 2021 Mar;80(3):312-320. doi: 10.1136/annrheumdis-2020-218870. Epub 2020 Dec 3. PMID 33272960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 123 sites in 16 countries (Belgium, Brazil, Canada, Chile, Czech Republic, France, Greece, Hungary, Italy, Japan, Netherlands, New Zealand, Portugal, Spain, United Kingdom, United States [including Puerto Rico]).
  Adults with active psoriatic arthritis (PsA) and a history of inadequate response or intolerance to at least one biologic disease modifying anti-rheumatic drug (bDMARD) were enrolled.
Pre-assignment Details: Participants were randomly assigned at a 1:1:2:2 ratio to one of four treatment groups below. Randomization was stratified by extent of psoriasis (≥ 3% body surface area [BSA] or < 3% BSA), current use of at least 1 DMARD, and number of prior failed biologic DMARDs (1 vs > 1), except for participants from Japan, for whom randomization was stratified by extent of psoriasis (≥ 3% BSA or < 3% BSA) only.
Groups:
- Placebo / Upadacitinib 15 mg: Participants randomized to receive placebo once daily up to week 24 followed by upadacitinib 15 mg once daily. All participants in Period 1 who were randomized to receive Placebo up to 24 weeks were pooled for the assessment of all outcome measures.
- Placebo / Upadacitinib 30 mg: Participants randomized to receive placebo once daily up to week 24 followed by upadacitinib 30 mg once daily. All participants in Period 1 who were randomized to receive Placebo up to 24 weeks were pooled for the assessment of all outcome measures. Participants in this group were switched to upadacitinib 15mg QD during Period 2 after week 116, following a protocol amendment.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily.
- Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily. Participants in this group were switched to upadacitinib 15mg QD during Period 2 after week 116, following a protocol amendment.
Period: Period 1
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 106 | 106 | 211 | 219
Received Study Drug | 106 | 106 | 211 | 218 (One randomized participant did not qualify per inclusion/exclusion criteria and discontinued prior to treatment.)
Completed Week 24 | 81 | 92 | 192 | 195
Completed (Completed Week 56 (Period 1)) | 69 | 77 | 167 | 166
Not Completed | 37 | 29 | 44 | 53
Not completed — Adverse Event | 7 | 7 | 12 | 14
Not completed — Withdrawal by Subject | 18 | 9 | 10 | 17
Not completed — Lost to Follow-up | 4 | 4 | 6 | 8
Not completed — Lack of Efficacy | 6 | 7 | 12 | 6
Not completed — Other | 2 | 2 | 4 | 7
Not completed — One participant did not qualify per inclusion/exclusion criteria and discontinued prior to treatment | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 69 | 77 | 167 | 165 (One participant who completed Period 1 did not enter Period 2.)
Switched to 15mg QD Upa Dosing in Period 2 (Participants receiving 30 mg once daily switched to 15 mg once daily during Period 2.) | 0 | 28 | 0 | 59
Completed | 55 | 55 | 131 | 126
Not Completed | 14 | 22 | 36 | 39
Not completed — Adverse Event | 4 | 7 | 10 | 10
Not completed — Withdrawal by Subject | 3 | 7 | 13 | 16
Not completed — Lost to Follow-up | 2 | 2 | 3 | 5
Not completed — Lack of Efficacy | 2 | 4 | 7 | 4
Not completed — COVID-19 Infection | 0 | 0 | 1 | 0
Not completed — Other | 3 | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo once daily for 24 weeks. This group includes all participants who went on to receive upadacitinib 15 mg or upadacitinib 30 mg after week 24.
- Upadacitinib 15 mg: Participants received upadacitinib 15 mg once daily for 24 weeks.
- Upadacitinib 30 mg: Participants received upadacitinib 30 mg once daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 212 | 211 | 218 | 641
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.53) | 53.0 (12.02) | 53.0 (11.94) | 53.4 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 113 | 115 | 348
  Male | 92 | 98 | 103 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 36 | 50 | 139
  Not Hispanic or Latino | 159 | 175 | 168 | 502
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 186 | 183 | 196 | 565
  Black or African American | 7 | 5 | 5 | 17
  American Indian/Alaska Native | 0 | 3 | 0 | 3
  Native Hawaiian or other Pacific Islander | 1 | 1 | 1 | 3
  Asian | 17 | 19 | 16 | 52
  Multiple | 1 | 0 | 0 | 1
Extent of Psoriasis [Count of Participants; unit: Participants] — The extent of psoriasis was measured by the physician as the total body surface area (BSA) involved with psoriasis. For purposes of clinical estimation, the total surface of the participant's palm and five digits was assumed to be approximately equivalent to 1% of BSA.
  Participants
    < 3% BSA | 81 | 81 | 87 | 249
    ≥ 3% BSA | 131 | 130 | 131 | 392
Number of Prior Failed Biologic DMARDs [Count of Participants; unit: Participants] — Failed treatment with prior biologic DMARD is defined as lack of efficacy after a minimum 12 week duration of therapy. The zero category includes participants with intolerance but not inadequate response to a biologic DMARD.
  Participants
    0 bDMARDS | 18 | 16 | 17 | 51
    1 bDMARD | 135 | 126 | 130 | 391
    2 bDMARDS | 35 | 35 | 46 | 116
    ≥ 3 bDMARDS | 24 | 34 | 25 | 83
Duration of Psoriatic Arthritis Symptoms [Mean (Standard Deviation); unit: years] | 14.6 (11.70) | 12.2 (8.81) | 13.3 (10.84) | 13.4 (10.54)
Duration of PsA Diagnosis [Mean (Standard Deviation); unit: years] | 11.0 (10.33) | 9.6 (8.36) | 9.7 (8.71) | 10.1 (9.18)
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  joints | 25.3 (17.62) | 24.9 (17.27) | 24.2 (15.87) | 24.8 (16.91)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  joints | 12.0 (8.85) | 11.3 (8.19) | 12.9 (9.41) | 12.1 (8.85)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a numeric rating scale (NRS) from 0 to 10. A score of 0 indicates "no pain" and a score of 10 indicates "worst possible pain." Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 209 | 208 | 218 | 635
    (all) | 6.6 (2.12) | 6.4 (2.13) | 6.2 (2.21) | 6.4 (2.16)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The participant was asked to rate their current psoriatic arthritis disease activity on a 0 to 10 NRS, where 0 indicates no disease activity and 10 indicates severe disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 209 | 208 | 218 | 635
    (all) | 6.8 (2.04) | 6.8 (1.91) | 6.7 (2.15) | 6.8 (2.04)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The physician rated the participant's current global psoriatic arthritis disease activity (independently from the participant's assessment) on a 0 to 10 NRS where 0 indicates no disease activity and 10 indicates severe disease activity.
  units on a scale | 6.5 (1.76) | 6.5 (1.80) | 6.6 (1.73) | 6.5 (1.76)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 209 | 208 | 218 | 635
    (all) | 1.23 (0.69) | 1.10 (0.61) | 1.19 (0.66) | 1.17 (0.66)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 10.40 (18.46) | 11.16 (18.55) | 10.53 (17.21) | 10.69 (18.05)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received placebo once daily for 24 weeks.
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 212 | 211 | 218
percentage of participants | 24.1 [18.3 to 29.8] | 56.9 [50.2 to 63.6] | 63.8 [57.4 to 70.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — The overall type I error rate of primary and ranked key secondary endpoints was strongly controlled using a graphical multiple testing procedure starting with the primary endpoint using α/2 for each dose followed by a prespecified α transfer path; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 32.8, 95% CI 2-sided [24.0 to 41.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 39.7, 95% CI 2-sided [31.1 to 48.3] — Response Rate Difference = Upadacitinib - Placebo

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 180 | 199 | 204
score on a scale | -0.10 [-0.16 to -0.03] | -0.30 [-0.37 to -0.24] | -0.41 [-0.47 to -0.35]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; MMRM analysis including treatment, visit, treatment-by-visit interaction, current DMARD use (yes/no) as fixed factors and Baseline value as covariate; Least Squares (LS) Mean Difference = -0.21, 95% CI 2-sided [-0.30 to -0.12] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.31, 95% CI 2-sided [-0.40 to -0.22] — Treatment Difference = Upadacitinib - Placebo

3. Secondary Outcome: Percentage of Participants Achieving a Static Investigator Global Assessment (sIGA) of Psoriasis of 0 or 1 and at Least a 2-point Improvement From Baseline (sIGA 0/1) at Week 16
Description: The sIGA is a 5 point scale ranging from 0 to 4, based on the investigator's assessment of the average elevation, erythema, and scaling of all psoriatic lesions at the current visit. A lower score indicates less severe psoriasis (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe).
Time Frame: Baseline and Week 16
Population: Full analysis set participants with a Baseline sIGA score ≥ 2; participants who prematurely discontinued from study drug prior to Week 16 or for whom sIGA data were missing at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 163 | 171 | 164
percentage of participants | 9.2 [4.8 to 13.6] | 36.8 [29.6 to 44.1] | 40.2 [32.7 to 47.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 27.6, 95% CI 2-sided [19.2 to 36.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 31.0, 95% CI 2-sided [22.3 to 39.8] — Response Rate Difference = Upadacitinib - Placebo

4. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 Response at Week 16
Description: PASI is a composite score based on the percentage of the body surface area (BSA) affected by psoriasis and the intensity of erythema (reddening), induration (thickening or hardening of the skin), and desquamation (peeling of the skin) of lesions assessed at 4 anatomic sites (head, upper extremities, trunk, and lower extremities). At each location, the percentage of BSA involvement is assigned a score from 0 (no involvement) to 6 (90% to 100% involvement), and erythema, induration, and desquamation are scored on a scale from 0 (no symptoms) to 4 (very marked).
  The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from Baseline in PASI score.
Time Frame: Baseline and Week 16
Population: Full analysis set participants with Baseline psoriasis BSA involvement ≥ 3%; participants who prematurely discontinued from study drug prior to Week 16 or for whom PASI data were missing at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 131 | 130 | 131
percentage of participants | 16.0 [9.7 to 22.3] | 52.3 [43.7 to 60.9] | 56.5 [48.0 to 65.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 36.3, 95% CI 2-sided [25.6 to 46.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 40.5, 95% CI 2-sided [29.9 to 51.0] — Response Rate Difference = Upadacitinib - Placebo

5. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 185 | 201 | 206
score on a scale | 1.62 [0.58 to 2.67] | 5.15 [4.14 to 6.15] | 7.06 [6.07 to 8.06]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 3.52, 95% CI 2-sided [2.07 to 4.98] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 5.44, 95% CI 2-sided [3.99 to 6.88] — Treatment Difference = Upadacitinib - Placebo

6. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 12
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue (e.g., I feel tired), functional fatigue (e.g., trouble finishing things), emotional fatigue (e.g., frustration), and social consequences of fatigue (e.g., limits social activity). Participants respond to the questions on a scale from 0 'not at all' to 4 'very much'. The FACIT Fatigue score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue subscale score ranges from 0 to 52, where higher scores represent less fatigue. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 184 | 201 | 206
score on a scale | 1.3 [0.1 to 2.5] | 5.0 [3.8 to 6.1] | 6.1 [4.9 to 7.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 3.7, 95% CI 2-sided [2.0 to 5.4] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; The overall type I error rate of primary and ranked key secondary endpoints was strongly controlled using a graphical multiple testing procedure starting with the primary endpoint using α/2 for each dose followed by a prespecified α transfer path; Test type: Superiority; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 4.8, 95% CI 2-sided [3.1 to 6.4] — Treatment Difference = Upadacitinib - Placebo

7. Secondary Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA) at Week 24
Description: A participant was classified as achieving MDA if 5 of the following 7 criteria were met:
  * Tender joint count (out of 68 joints) ≤ 1
  * Swollen joint count (out of 66 joints) ≤ 1
  * PASI score ≤ 1 (score ranges from 0 - 72) or percent BSA involved with psoriasis ≤ 3%
  * Patient's assessment of pain ≤ 1.5 (NRS from 0 to 10)
  * Patient's Global Assessment of disease activity ≤ 2 (NRS from 0 to 10)
  * HAQ-DI score ≤ 0.5 (index score ranges from 0 to 3)
  * Leeds Enthesitis Index ≤ 1 (assesses the presence or absence of enthesitis at 3 bilateral sites, with an overall score range from 0 to 6)
Time Frame: Week 24
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 24 or for whom data were missing at Week 24, or who met rescue criteria at Week 16 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 212 | 211 | 218
percentage of participants | 2.8 [0.6 to 5.1] | 25.1 [19.3 to 31.0] | 28.9 [22.9 to 34.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 22.3, 95% CI 2-sided [16.0 to 28.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 26.1, 95% CI 2-sided [19.7 to 32.5] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Change From Baseline in Self-Assessment of Psoriasis Symptoms (SAPS) Score at Week 16
Description: The SAPS is an 11-item self-assessment of psoriasis symptoms that includes questions on: pain, itching, redness, scaling, flaking, bleeding, burning, stinging, tenderness, pain due to skin cracking, and joint pain. Each item is scored from 0 to 10, with 0 being least severe and 10 being most severe. The total score is generated by summing the 11 items and ranges from 0 to 110 (worst). A negative change from Baseline in the total score indicates improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 16 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 182 | 191 | 200
score on a scale | -1.5 [-4.7 to 1.8] | -24.4 [-27.5 to -21.2] | -29.7 [-32.8 to -26.6]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -22.9, 95% CI 2-sided [-27.4 to -18.4] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -28.2, 95% CI 2-sided [-32.7 to -23.8] — Treatment Difference = Upadacitinib - Placebo

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 212 | 211 | 218
percentage of participants | 4.7 [1.9 to 7.6] | 31.8 [25.5 to 38.0] | 37.6 [31.2 to 44.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 27.0, 95% CI 2-sided [20.1 to 33.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 32.9, 95% CI 2-sided [25.9 to 39.9] — Response Rate Difference = Upadacitinib - Placebo

10. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 212 | 211 | 218
percentage of participants | 0.5 [0.0 to 1.4] | 8.5 [4.8 to 12.3] | 16.5 [11.6 to 21.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 8.1, 95% CI 2-sided [4.2 to 11.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 16.0, 95% CI 2-sided [11.0 to 21.1] — Response Rate Difference = Upadacitinib - Placebo

11. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 2
Description: as for outcome 1
Time Frame: Baseline and Week 2
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 2 or for whom ACR data were missing at Week 2 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 212 | 211 | 218
percentage of participants | 10.8 [6.7 to 15.0] | 32.7 [26.4 to 39.0] | 33.5 [27.2 to 39.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 21.9, 95% CI 2-sided [14.3 to 29.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for the main stratification factor of current DMARD use (yes/no); Response Rate Difference = 22.6, 95% CI 2-sided [15.1 to 30.2] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment to the end of the study. For Period 1, the median time participants were followed was: 414 days (15mg Upa); 413 days (30mg Upa); 190 days (Pooled Placebo ICF to week 24); 415 days (Pbo 15mg Upa); and 415 days (Pbo 30mg Upa). For Period 2, the median time participants were followed was: 712 days (15mg Upa); 701 days (30mg Upa); 703 days (Pbo 15mg Upa); 672 days (Pbo 30mg Upa); and 223 days (Switched to 15mg Upa).
Description: Participants receiving Upadacitinib 30 mg once daily were switched to Upadacitinib 15 mg once daily during Period 2. Following the switch, adverse events were pooled for these participants to end-of-study (EOS).
Groups:
- Period 1: Upadacitinib 15 mg (ICF to Week 56): Participants randomized to receive Upadacitinib 15 mg once daily to Week 56.
- Period 1: Upadacitinib 30 mg (ICF to Week 56): Participants randomized to receive Upadacitinib 30 mg once daily to Week 56.
- Period 1: Pooled Placebo (ICF to Week 24): This group includes all participants in Period 1 who were randomized to receive Placebo once daily to Week 24.
- Period 1: Placebo / Upadacitinib 15 mg (Week 24 to Week 56): Participants were randomized to receive placebo once daily for 24 weeks followed by upadacitinib 15 mg once daily to Week 56. AEs in this group were reported while participants received 15 mg upadacitinib from Week 24 to Week 56.
- Period 1: Placebo / Upadacitinib 30 mg (Week 24 to Week 56): Participants were randomized to receive placebo once daily for 24 weeks followed by upadacitinib 30 mg once daily to Week 56. AEs in this group were reported while participants received 30 mg upadacitinib from Week 24 to Week 56.
- Period 2: Upadacitinib 15 mg (Week 56 to EOS): Participants randomized to receive upadacitinib 15 mg once daily in Period 2 from Week 56 to EOS.
- Period 2: Upadacitinib 30 mg (Week 56 to EOS): Participants randomized to receive upadacitinib 30 mg once daily in Period 2 from Week 56 to EOS. Participants in this group were switched to upadacitinib 15 mg once daily during Period 2 after week 116, following a protocol amendment.
- Period 2: Placebo / Upadacitinib 15 mg (Week 56 to Week EOS): Participants from the Period 1 Placebo / Upadacitinib 15 mg group received 15 mg upadacitinib once daily from Week 56 to EOS.
- Period 2: Placebo / Upadacitinib 30 mg (Week 56 to EOS): Participants from the Period 1 Placebo / Upadacitinib 30 mg group were to receive 30 mg upadacitinib once daily from Week 56 to EOS. Participants in this group were switched to upadacitinib 15 mg once daily during Period 2 after week 116, following a protocol amendment.
- Period 2: Pooled Upadacitinib Groups Who Switched From 30 mg to 15 mg in Period 2: All participants in Period 2 who switched from 30 mg to 15 mg upadacitinib to EOS during Period 2. This group includes all participants who received any upadacitinib 30 mg in Period 2 and switched dose to upadacitinib 15 mg once daily during Period 2 (following a protocol amendment, after week 116). The AEs in this group were reported while participants received 15 mg upadacitinib once daily.
Arm/Group | Period 1: Upadacitinib 15 mg (ICF to Week 56) | Period 1: Upadacitinib 30 mg (ICF to Week 56) | Period 1: Pooled Placebo (ICF to Week 24) | Period 1: Placebo / Upadacitinib 15 mg (Week 24 to Week 56) | Period 1: Placebo / Upadacitinib 30 mg (Week 24 to Week 56) | Period 2: Upadacitinib 15 mg (Week 56 to EOS) | Period 2: Upadacitinib 30 mg (Week 56 to EOS) | Period 2: Placebo / Upadacitinib 15 mg (Week 56 to Week EOS) | Period 2: Placebo / Upadacitinib 30 mg (Week 56 to EOS) | Period 2: Pooled Upadacitinib Groups Who Switched From 30 mg to 15 mg in Period 2
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/219 | 1/212 | 0/79 | 0/90 | 5/167 | 0/165 | 0/69 | 2/77 | 0/87
Serious Adverse Events (participants affected / at risk) | 22/211 | 25/219 | 5/212 | 3/79 | 6/90 | 24/167 | 19/165 | 7/69 | 12/77 | 5/87
Other Adverse Events (participants affected / at risk) | 111/211 | 139/219 | 87/212 | 32/79 | 34/90 | 111/167 | 99/165 | 42/69 | 49/77 | 34/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Upadacitinib 15 mg (ICF to Week 56) (N=211) | Period 1: Upadacitinib 30 mg (ICF to Week 56) (N=219) | Period 1: Pooled Placebo (ICF to Week 24) (N=212) | Period 1: Placebo / Upadacitinib 15 mg (Week 24 to Week 56) (N=79) | Period 1: Placebo / Upadacitinib 30 mg (Week 24 to Week 56) (N=90) | Period 2: Upadacitinib 15 mg (Week 56 to EOS) (N=167) | Period 2: Upadacitinib 30 mg (Week 56 to EOS) (N=165) | Period 2: Placebo / Upadacitinib 15 mg (Week 56 to Week EOS) (N=69) | Period 2: Placebo / Upadacitinib 30 mg (Week 56 to EOS) (N=77) | Period 2: Pooled Upadacitinib Groups Who Switched From 30 mg to 15 mg in Period 2 (N=87)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GOITRE (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINE ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BURSITIS INFECTIVE STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EXTRADURAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIV INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC HAEMOTHORAX (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RAPIDLY PROGRESSIVE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTRADUCTAL PAPILLARY BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN THECA CELL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CAROTID ARTERY INSUFFICIENCY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPEECH DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Upadacitinib 15 mg (ICF to Week 56) (N=211) | Period 1: Upadacitinib 30 mg (ICF to Week 56) (N=219) | Period 1: Pooled Placebo (ICF to Week 24) (N=212) | Period 1: Placebo / Upadacitinib 15 mg (Week 24 to Week 56) (N=79) | Period 1: Placebo / Upadacitinib 30 mg (Week 24 to Week 56) (N=90) | Period 2: Upadacitinib 15 mg (Week 56 to EOS) (N=167) | Period 2: Upadacitinib 30 mg (Week 56 to EOS) (N=165) | Period 2: Placebo / Upadacitinib 15 mg (Week 56 to Week EOS) (N=69) | Period 2: Placebo / Upadacitinib 30 mg (Week 56 to EOS) (N=77) | Period 2: Pooled Upadacitinib Groups Who Switched From 30 mg to 15 mg in Period 2 (N=87)
DIARRHOEA (Gastrointestinal disorders) | 8 (8) | 15 (18) | 12 (13) | 3 (4) | 3 (3) | 5 (5) | 3 (5) | 1 (1) | 2 (2) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 8 (8) | 12 (12) | 7 (8) | 0 (0) | 1 (1) | 4 (5) | 10 (10) | 0 (0) | 0 (0) | 1 (1)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 1 (1) | 5 (5) | 1 (1)
BRONCHITIS (Infections and infestations) | 17 (20) | 15 (16) | 5 (5) | 5 (7) | 4 (4) | 15 (17) | 8 (10) | 6 (6) | 4 (5) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 21 (21) | 12 (12) | 7 (7) | 7 (7) | 14 (17)
HERPES ZOSTER (Infections and infestations) | 8 (8) | 13 (13) | 2 (2) | 2 (2) | 5 (5) | 10 (10) | 13 (13) | 3 (3) | 5 (5) | 1 (1)
INFLUENZA (Infections and infestations) | 14 (16) | 13 (14) | 3 (3) | 2 (2) | 2 (3) | 3 (4) | 6 (6) | 2 (2) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 24 (29) | 29 (34) | 17 (18) | 5 (5) | 6 (8) | 14 (17) | 12 (13) | 7 (8) | 6 (6) | 5 (6)
PNEUMONIA (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 4 (6) | 1 (1)
SINUSITIS (Infections and infestations) | 8 (9) | 9 (10) | 9 (11) | 3 (4) | 2 (2) | 7 (9) | 7 (7) | 2 (4) | 6 (8) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 22 (27) | 29 (34) | 10 (13) | 6 (7) | 2 (2) | 15 (15) | 9 (13) | 5 (5) | 6 (7) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 19 (24) | 16 (18) | 12 (14) | 4 (4) | 4 (4) | 17 (24) | 14 (22) | 8 (11) | 9 (12) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5) | 11 (13) | 1 (1) | 0 (0) | 4 (4) | 6 (7) | 6 (6) | 3 (3) | 2 (2) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 9 (10) | 22 (29) | 4 (4) | 2 (3) | 4 (5) | 13 (15) | 9 (9) | 5 (5) | 6 (7) | 2 (2)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 0 (0)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 13 (14) | 7 (8) | 11 (12) | 2 (2) | 3 (3) | 12 (15) | 16 (18) | 9 (9) | 8 (8) | 8 (8)
HYPERTENSION (Vascular disorders) | 8 (9) | 10 (10) | 10 (12) | 4 (4) | 3 (3) | 19 (20) | 11 (11) | 5 (5) | 7 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT03104374/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03104374/SAP_003.pdf